CLINICAL TRIAL: NCT07192718
Title: A Pilot Feasibility Trial for a Comprehensive Multimodal Intervention to Assess Global Recovery Following Cesarean Delivery
Brief Title: Using Empowered Relief and Education To Help Postpartum Women Recover After Cesarean Delivery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, PSultan, Professor of Anesthesiology, Perioperative and Pain Medicine (Obstetrics), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80489; 5R90HD118650 (NIH)
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cesarean Section Complications; Postpartum Care
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-Session pain relief skills session (Empowered Relief) and Education (Experimental): Participants will view educational content online on postpartum care and attend a 2 hour Empowered Relief session at the beginning of the study period.
  Standard of care will be maintained for all participants, and supplemented with Educational content and Empowered Relief.
  Interventions: Behavioral: Empowered Relief; Other: Education
- Standard of Care (No Intervention): Participants will follow their current standard of care.

INTERVENTIONS:
Behavioral: Empowered Relief — The participants will attend a pain relief skills intervention (Empowered Relief). The two-hour session is delivered by a certified instructor and includes pain neuroscience education, 3 core pain management skills, experiential exercises, completion of a personalized plan for empowered relief. Participants download a binaural relaxation audio file for daily use.
  Other Names: 1-Session Pain Relief Skills Intervention
  Arms: 1-Session pain relief skills session (Empowered Relief) and Education
Other: Education — Educational content: Participants view videos online focusing on specific areas of postpartum recovery (Sleep, Mental Health, Physical Therapy, Obstetric care).
  Arms: 1-Session pain relief skills session (Empowered Relief) and Education

SUMMARY:
The purpose of this study is to study the effect of a pain relief skills session (Empowered Relief) and educational content on global postpartum recovery at 12 weeks post cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years of age or older
* Any woman scheduled for a cesarean delivery in the Stanford Healthcare system with a viable birth
* English fluency
* Ability to adhere to and complete study protocols
* Access to smart device for zoom / video meetings

Exclusion Criteria:

* <18yrs
* chronic pain prior to pregnancy
* Cognitive impairment, non-English speaking, or psychological factors that would preclude comprehension of material and/or full participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants registering for Empowered Relief session | Baseline (up to 2 weeks)
Percentage of participants attending Empowered Relief session | Treatment (up to 2 weeks)
Empowered Relief: Participant Satisfaction Scale Score | 1 - 2 weeks Post treatment
  Participant satisfaction will be measured using a 7 item questionnaire (scale ranges from 0 - 42, higher ratings represent greater satisfaction with the treatment).
Empowered Relief: Participant Treatment Skills Use Scale Score | Week 3, Week 8, Week 14
  Participant treatment skills use will be measured with a 5 items questionnaire (scale ranges from 0 - 25, higher ratings represent increased time using treatment).
Percentage of participants watching educational content | Treatment (up to 2 weeks), Week 3
Educational content: Participant Satisfaction Scale Score | 1 - 2 weeks Post treatment, Week 3, Week 8, Week 14
  Participant satisfaction will be measured using a 7 item questionnaire with three scored items: overall usefulness (0-6), the usefulness rating of each module (0-6), and frequency of use (0-3). The composite score ranges from 0-15, with higher scores indicating greater satisfaction and use. Additional checklist and free-text items capture engagement but are not included in the score.

SECONDARY OUTCOMES:
Change from baseline in PROMIS Pain Interference 8a scale score | Baseline, Week 3, Week 8, Week 14
  Participants complete Patient Reported Outcomes Measurement Outcomes System (PROMIS) Pain Interference 8a questionnaire, an 8-item scale assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days. (Score range 8 - 40, higher scores represent a greater degree of pain interference).
Change from baseline in PROMIS Pain Intensity 3a scale score | Baseline, Week 3, Week 8, Week 14
  Participants complete PROMIS Pain Intensity 3a questionnaire, a 3-item scale assessing average pain intensity for the past 7 days. (Score range 3 - 15, higher score represents a greater degree of pain intensity)
Change from baseline in Pain Catastrophizing Scale Score | Baseline, Week 3, Week 8, Week 14
  Participants complete Pain Catastrophizing questionnaire, a 13-item scale assessing an individual's pain experience (Score range 0 - 52, higher score represents a greater degree of pain catastrophizing)
Change from baseline in Pain Interference Scale Score via SMS | Baseline through end of study (up to 14 weeks)
  Participants complete twice weekly questionnaire to assess pain interference via SMS. (Score range 0 - 10, higher score represents a greater degree of interference)
Response rate to Pain Interference scale score via SMS | Baseline through end of study (up to 14 weeks)
  This outcome determines the percentage of participants responding to the twice weekly pain interference scale score via SMS text.
Change from baseline in PROMIS Sleep Disturbance 8a scale score | Baseline, Week 3, Week 8, Week 14
  Participants complete Patient Reported Outcomes Measurement Outcomes System (PROMIS) Sleep Disturbance 8a questionnaire, an 8-item scale assessing self-reported perceptions of sleep quality, sleep depth, restoration, perceived difficulties and concerns with getting to sleep/staying asleep, as well as perceptions of the adequacy and satisfaction with sleep over the past 7 days. (Score range 8 - 40, higher scores represent a greater degree of sleep disturbance).
Change from baseline in STanford Obstetric Recovery checKlist (STORK) scale score | Baseline, Week 2, Week 3, Week 8, Week 14
  Participants complete the STORK questionnaire, a 47-item scale assessing postpartum recovery over the past 7 days. (Score range 0 - 188, higher score represents a greater degree of recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Pervez Sultan, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Wish whom? Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. For what types of analysis? For individual participant data meta-analysis By what mechanism will data be made available? Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be provided).

REFERENCES:
- [Background] Ciechanowicz S, Joy RR, Kasmirski J, Blake L, Carvalho B, Sultan P. Incidence, Severity, and Interference of Chronic Postsurgical Pain After Cesarean Delivery: A Systematic Review and Meta-analysis. J Clin Anesth. 2025 Jun;104:111832. doi: 10.1016/j.jclinane.2025.111832. Epub 2025 Apr 24. PMID 40279839
- [Background] Sultan P, Pandal P, Murthy A, Guo N, Farber MK, Toledo P, Higgins N, Fiore JF Jr, Domingue BW, Khorasani E, Jensen SE, Lyell DJ, Carvalho B; Stanford Obstetric Recovery Checklist (STORK) Investigators. Development and Validation of the Stanford Obstetric Recovery Checklist (STORK): A Delphi Consensus and Multicenter Clinical Validation Study. JAMA Netw Open. 2025 Apr 1;8(4):e255713. doi: 10.1001/jamanetworkopen.2025.5713. PMID 40244582